CLINICAL TRIAL: NCT02552628
Title: DEEP BRAIN STIMULATION FOR SEVERE DYSTONIA ASSOCIATED WITH WILSON'S DISEASE. A Prospective Multicenter Meta-analysis of Nof1 Trials
Brief Title: WILSTIM - DBS (WILson STIMulation - Deep Brain Stimulation)
Acronym: WILSTIM DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL14_0448; IDRCB (Other: 2015-A00211-48)
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2023-06

CONDITIONS: Severe Dystonia; Wilson's Disease
Keywords: Wilson's Disease; Deep Brain Stimulation; dystonia
MeSH Terms: conditions — Dystonia; Hepatolenticular Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulation "on" (Experimental): The deep brain stimulation is "on"
  Interventions: Device: Medtronic, Activa® PC "on"
- Stimulation "off" (Sham Comparator): The deep brain stimulation is "off"
  Interventions: Device: Medtronic, Activa® PC "off"

INTERVENTIONS:
Device: Medtronic, Activa® PC "on"
  Arms: Stimulation "on"
Device: Medtronic, Activa® PC "off"
  Arms: Stimulation "off"

SUMMARY:
Dystonia in Wilson's disease represent a major issue. The persistence of disabling motor symptoms despite medical treatments justifies conducting a study on deep brain stimulation (DBS) in Wilson's disease (WD). For bradykinetic patients, subthalamic nucleus (STN) could be considered as a better target than the globus pallidus (GPi). For patients with hyperkinetic dystonia, the internal globus pallidus (GPi) will be chosen as the target of DBS.

The investigators hypothesize that STN DBS will improve Wilson's disease patients, who, despite copper chelators drugs, are still impaired by severe dystonia and akinesia (more or less associated with other movement disorders).

The investigators primary objective is to demonstrate the efficacy of STN/GPi DBS on dystonia associated with Wilson's disease.

Secondary objectives:

* To evaluate the impact of STN/GPi DBS on other movements disorders (tremor, Parkinsonism, chorea) observed in Wilson's disease.
* To describe cognitive status of patients and to evaluate the consequences of STN/GPi DBS on cognition and behavioral aspects of the disease.
* To evaluate the consequences of the stimulation on speech and swallowing.
* To evaluate the social impact of STN/GPi DBS in Wilson's disease.
* To evaluate the safety of STN/GPi DBS in the specific context of Wilson's disease.

DETAILED DESCRIPTION:
4 periods of stimulation on and off, sequence randomized at Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 60 years.
* Severe neurological form of Wilson's disease with predominant dystonia and akinetic-rigid syndrome, despite optimized treatment stabilized for at least 6 months.
* Important disability due to abnormal movements (Rankin score=2 to 4).
* Absence of dementia (MMS > 24 and BREF > 15).
* Stable psychiatric status and absence of severe depression (BDI <28).
* Social security coverage.
* Signature of informed consent. (signature of legal guardian for subjects under protection)

Exclusion Criteria:

* Severe hepatopathy with coagulation disorders (Platelet count < 100 G / l; INR > 1.5; V factor deficit; low level of fibrinogen < 1g/dL; increased of fibrin degradation products; low level of antithrombin).
* Liver transplanted patients < 2 years
* Patients under immunosupressive drugs and corticoids regimen.
* Participation to another biomedical research involving any drugs.
* Severe and uncontrolled psychosis or depression.
* Major atrophy on brain MRI that could represent a problem for leads implantation.
* Necrosis of the STN/GPi on brain MRI.
* Female subjects who are pregnant or lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in movement disorder evaluated by the Canadian Occupational Performance Measure (COPM) performance and satisfaction scores | 21 months
  Efficacy will be assessed by the change in the COPM performance and satisfaction scores after each 4 month-period of stimulation on and off, using blinded evaluations. The COPM is a standardized outcome measure widely used in occupational therapy. This tool can facilitate the identification of functional difficulties and individualized subject-specific priorities for intervention, which may not be captured with other standardized scales.

SECONDARY OUTCOMES:
Other movement disorder will be assessed by the reduction of the Burke-Fahn-Marsden (BFM) dystonia scale score | 21 months
  The reduction of the Burke-Fahn-Marsden (BFM) dystonia scale score is evaluated after each 4 month-period of stimulation on and off, using blinded video evaluations. This scale is the standard of assessments on dystonia and Parkinson.
Change in other movement disorder evaluated by the Clinical global impression (CGI) scale | 21 months
Change in other movement disorder evaluated by the Unified Wilson Disease Rate Scale (UWDRS) | 21 months
  The UWDRS consists of 3 sections, including: consciousness, a historical review based on the Barthel scale, and neurological examination.
Cognitive evaluation using the Mini Mental Status Examination (MMSE) | Screening visit (2 days)
  The MMSE is a brief 30-point questionnaire test commonly used to screen for dementia.
Cognitive evaluation using the Frontal Assessment Battery (FAB) | Screening visit (2 days)
  The FAB is a brief tool used to assess dysexecutive symptoms.
Cognitive evaluation using the BDI-II (Beck Depression Inventory) | Screening visit (2 days)
  The BDI-II is a self- report inventory for measuring the severity of depression.
Cognitive evaluation using the similarities and matrix reasoning tests from the Wechsler Adult Intelligence Scale (WAIS-IV) | Pre-surgery visit (2 days)
  The test of similarities measures concrete, functional, and abstract concept formation. The test of matrix reasoning measures nonverbal analytical reasoning.
Cognitive evaluation using the Modified Card Sorting Test (MCST) | Pre-surgery visit (2 days)
  The MCST assess problem solving and the ability to shift cognitive strategies in response to changing environmental contingencies.
Cognitive evaluation using the Trail Making Test (TMT) | Pre-surgery visit (2 days)
  The TMT assess visuo-motor speed and task switching abilities.
Cognitive evaluation using the phonemic verbal fluency task | Pre-surgery visit (2 days)
  The phonemic verbal fluency task assesses intrinsic response generation.
Cognitive evaluation using the 16-items free and cued recall test (RL/RI 16-items) | Pre-surgery visit (2 days)
  The RL/RI 16-items test assesses episodic memory and especially abilities to retrieve information from memory.
Change in cognitive outcome evaluated by the Tasks of the test of Attentional Performance (TAP) | 21 months
  The TAP is a normalized computerized battery to assess attentional and executive abilities.
Change in behavioral and neuropsychiatric outcome evaluated by the "Inventaire du Syndrome Dysexécutif Comportemental" (ISDC) | 21 months
  The ISDC assesses behavioral dysexecutive symptoms.
Change in behavioral and neuropsychiatric outcome evaluated by the Brief Psychiatric Rating Scale with anchor (BPRS-E(A)) | 21 months
  The BPRS-E(A) is widely used to measure psychiatric symptoms and unusual behavior.
Change in dysarthria and deglutition outcome evaluated by the spontaneous speech and reading | 21 months
Change in dysarthria and deglutition outcome evaluated by the the "Batterie d'Evaluation de la Dysarthrie" (BECD) | 21 months
  This BECD score provides a global assessment of dysarthria severity.
Change in dysarthria and deglutition outcome evaluated by the Voice Handicap Index (VHI) | 21 months
  The VHI is a questionnaire to quantify the functional, physical and emotional impacts of a voice disorder on a patient's quality of life.
Change in dysarthria and deglutition outcome evaluated by the maximum phonation time | 21 months
Change in dysarthria and deglutition outcome evaluated by the GRBAS (Grade, Roughness, Breathiness, Asthenia, Strain) scale | 21 months
  Auditory-perceptual evaluation method for hoarseness is the GRBAS scale of the Japan Society of Logopedics and Phoniatrics, which rates hoarseness.
Change in dysarthria and deglutition outcome evaluated by the Deglutition Handicap Index (DHI) | 21 months
  The DHI questionnaire is composed of statements on deglutition related aspects in daily life. It is subdivided in three domains: physical (S) (symptoms related to swallowing), functional (F) (nutritional and respiratory consequences) and emotional (E) (psychosocial consequences).
Change in dysarthria and deglutition outcome evaluated by the timed test of swallowing capacity | 21 months
Change in social outcome evaluated by the Zarit Burden Inventory (ZBI) | 21 months
  The ZBI is a popular caregiver self-report measure used by many aging agencies.
Tolerance of Deep Brain Stimulation: occurrence of serious adverse events | 23 months
  Clinical examination focusing specifically on vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane THOBOIS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hospices Civils de Lyon, Lyon
  - Hopital Lariboisiere, Paris
  - Hôpital Fondation Adolphe de Rothschild Paris, Paris

REFERENCES:
- [Result] Laurencin C, Poujois A, Bonjour M, Demily C, Klinger H, Roze E, Leclert V, Danaila T, Langlois-Jacques C, Couchonnal E, Woimant F, Obadia MA, Perez G, Pernon M, Blanchet L, Broussolle E, Vidailhet M, Kassai B, Moro E, Karachi C, Polo G, Grabli D, Portefaix A, Thobois S. Deep brain stimulation for severe dystonia associated with Wilson disease: A prospective multicenter meta-analysis of an N-of-1 trial. Eur J Neurol. 2025 Jan;32(1):e16524. doi: 10.1111/ene.16524. Epub 2024 Oct 29. PMID 39468897